CLINICAL TRIAL: NCT05259319
Title: An Open-label, Multi-centric, Phase I, Evaluating the Safety and the Efficacy of Combination of Atezolizumab, Tiragolumab and and Stereotactic Body Radiation Therapy in Patients With Oligometastatic Multiorgan (IMMUNOs-SBRT)
Brief Title: Study Evaluating the Safety and the Efficacy of Combination of Atezolizumab, Tiragolumab and and Stereotactic Body Radiation Therapy in Patients With Oligometastatic Multiorgan (IMMUNOs-SBRT)
Acronym: IMMUNOs-SBRT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-003848-25
Record Dates: First submitted 2022-01-24; First posted 2022-02-28 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Non Small Cell Lung Cancer; Metastatic Bladder Cancer; Metastatic Renal Cell Carcinoma; Metastatic Head and Neck Cancer
Keywords: Atezolizumab; Tiragolumab; Cancer; Stereotactic body radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Head and Neck Neoplasms; Neoplasms | interventions — atezolizumab; Tiragolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Tiragolumab + SBRT (Experimental): Atezolizumab + Tiragolumab (every 21 days during 24 months or until progression) + SBRT (treatment will be delivered on 5 days).
  The combination of SBRT and Immunotherapies will be performed using to different schemes. For the 6 first inclusions the combination will use a sequential scheme. If the safety criteria are respected the following patients will be able to be treated by concomitant scheme.
  Interventions: Drug: Atezolizumab 60 MG/1 ML Intravenous Solution [TECENTRIQ]; Drug: Tiragolumab; Radiation: Stereotactic body radiation therapy (SBRT)

INTERVENTIONS:
Drug: Atezolizumab 60 MG/1 ML Intravenous Solution [TECENTRIQ] — Treatment given every 21 days during 24 months or until progression
Drug: Tiragolumab — Treatment given every 21 days during 24 months or until progression
Radiation: Stereotactic body radiation therapy (SBRT) — Radiothérapy is delivered as a hypofractionated schedule of 3 doses of 8Gy (idealy on Monday, Wednesday and Friday, or 3 sessions over a week, respecting at least 24 hours between each fraction)

SUMMARY:
This study (phase I clinical trial and expansion cohorts) will evaluate safety and efficacy of combination of atezolizumab and tiragolumab, with concomitant or sequential SBRT for four oligometastatic cancer cohorts. This study will allow to developpe one or several randomized Phase II clinical trials for the more promising indications

DETAILED DESCRIPTION:
This study will be composed of 2 stepms. First step will be a phase I with the aim to establish the recommended safety scheme of administration (concomitant or sequential) of tiragolumab + atezolizumab + SBRT. The phase I will enrolled only patients from the cohort 1 (metastatic non-small cell lung cancer).

The second step will be an expansion cohorts phase at the recommended scheme of administration. The second step will enrolled patients from 4 different cohorts (metastatic non-small cell lung cancer, metastatic bladder cancer, metastatic renal cell carcinoma, metastatic head and neck carcinoma).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* ECOG, Performance status ≤ 1,
* Minimum 3 measurable lesions, with at least one lesion which cannot be irradiated for testing the abscopal effect and at least 2 irradiable lesions.
* Life expectancy > 6 months,
* At least one non irradiated tumor site that can be biopsied for research purpose,
* Participant must have following advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement:

Cohort 1 : patient with metastatic non small lung cancer / tumor without oncogenic addiction (EGFR/ALK/ROS/BRAF) which progress after platin based chemotherapy and immunotherapy given as sequential or concomitant therapy.

Cohort 2 : Bladder cancer / Patient with progression following platin based therapy or without maintenance with anti PD1/PD-L1. Patient have to recieve Enfortumab Vedotin before inclusion if the treatment is available. Unless indication by the investigator Cohort 3 : Renal cell carcinoma / Second-line therapy after an anti-angiogenic plus immunotherapy or immunotherapy.

Cohort 4 : Head and neck carcinoma / First line locoregional or metastatic recurrence

* Participants who received prior anti-PD-1/L1 therapy must fulfill the following requirements Have achieved a complete response, partial response or stable disease and subsequently had disease progression while still on anti-PD-1/L1 therapy Have received at least two doses of an approved anti-PD-1/L1 therapy (by any regulatory authority)
* Adequate hematological, renal, metabolic and hepatic functions:

Hemoglobin ≥ 9 g/dl (participants may have received prior red blood cell [RBC] transfusion, if clinically indicated); absolute neutrophil count (ANC) ≥ 1.5 G/l, platelet count ≥ 100 G/l, white blood cell count ≥ 2.5 G/l (or within local laboratory normal limits) and lymphocyte count ≥ 0.75 G/l Alkaline phosphatase (AP), alanine aminotransferase (ALT) and aspartate aminotransferase (ASP) ≤ 2.5 x upper limit of normality (ULN) (≤ 5 x ULN in case of extensive skeletal involvement for AP exclusively and ≤ 5 x ULN in case of liver metastasis for AST and ALT).

Total bilirubin ≤ 1.5 x ULN, (3 x ULN for gilbert disease) Albumin ≥ 25 g/l. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance (CrCl) ≥ 30 ml/min (according to Cockcroft and Gault formula).

INR ≤ 1.5 x ULN aPTT ≤ 1.5 X ULN Serum calcium within normal laboratory ranges,

* No prior or concurrent malignant disease if more recent than 3 years
* At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy

Criteria to confirm inclusion:

* At least 2 mesurable lesions should be able to receveid 3 X 8 Gy by SBRT according to the dose constraints to organs at risk (OAR) imposed by the protocol
* In case of lesion previously treated by radiotherapy, the constraints on the organs at risk must be respected after having summed up the treatment plans.
* Confirmation of 3 measureable lesions, with at least one lesion which cannot be irradiated for testing the abscopal effect and at least 2 irradiable lesions. Those lesions must be uni-dimensionally ≥ 10 mm considered as measurable according to RECIST v1.1

Exclusion Criteria:

* Evidence of symptomatic central nervous system (CNS) or leptomeningeal metastases,
* Women who are pregnant or breast feeding,
* Participation in a study involving a medical or therapeutic intervention in the last 30 days from first treatment administration,
* Previous enrolment in the present study,
* Participant unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons,
* Known hypersensitivity to any involved study drug or of its formulation components,
* History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins,
* Treatment with systemic immunosuppressive medications including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents within 2 weeks prior to inclusion. Systemic corticosteroids is not allowed but at physiologic doses meaning less than 10 mg/day of prednisone or its equivalent. The use of inhaled corticosteroids and mineral corticoids is allowed.
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days before pre inclusion,
* Any of the following cardiac criteria:

Congestive heart failure ≥ New York Heart Association (NYHA) class 2,

* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), Myocardial infarction less than 6 months before pre-inclusion Uncontrolled cardiac arrhythmias, Known left ventricular ejection fraction (LVEF) <50%
* Individuals deprived of liberty or placed under legal guardianship, curatorship or judicial protection.
* Prior organ transplantation, including allogeneic stem cell transplantation,
* Known clinically significant liver disease, including, alcoholic, or other hepatitis, cirrhosis, fatty liver and inherited liver disease, active viral with positive viralDNA detection.
* History of intra-abdominal inflammatory process within the last 12 months such as, but not limited to, diverticulitis, peptic ulcer disease or colitis.
* History of autoimmune disease including, but not limited to systemic lupus erythematosus (SLE), Sjögren's syndrome, glomerulonephritis, multiple sclerosis, rheumatoid arthritis, vasculitis, systemic immune activation, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Guillain-Barré syndrome, Bell's palsy.

Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible, Participants with controlled Type I diabetes mellitus on a stable insulin regimen are eligible, Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with only dermatologic manifestations <10% of the skin (e.g., participants with psoriatic arthritis would be excluded) are eligible.

* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Poorly controlled Type II diabetes mellitus defined as a screening fasting plasma glucose ≥160 mg/dL (or 8.8 mmol/L).
* Severe infections within 2 weeks prior to inclusion, including but not limited to SARS-Cov-2 infection, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Received therapeutic oral or IV antibiotics within 2 weeks prior to pre-inclusion. Participants receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Any contraindication to tumor biopsy,
* Participant with spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >2 weeks prior to pre-inclusion.
* Administration of a live, attenuated vaccine within 4 weeks before the start of study medication or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination is allowed during influenza season only (approximatively October to March).
* Patient with a known history of Human Immunodeficiency Virus (HIV) (HIV1/2 antibodies) or known acquired immunodeficiency syndrome (AIDS),
* Patients with EBV infection (Positive EBV viral capsid antigen IgM test at screening)
* Active tuberculosis
* Concomitant use of prohibited concomitant therapy (cf paragraph 6.5.2.2) or anticipation that such concomitant medication/therapies will be required during the study
* For NSCLC indication, patients with lymphoepithelioma-like carcinoma are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Phase I : to evaluate safety of SBRT | The first 5 weeks (35 days) after the first dose of study treatment for sequential administration (3X8 Gy of radiotherapy and 3 dosing of immunotherapy)
  Using the following DLTs (DLT are defined by the following events related to study treatments (SBRT and/or tiragolumab, atezolizumab) :
  * grade 3 pneumopathy (except if return to grade ≤2 within 7 days)
  * grade 3 radiation dermatitis (except if return to grade ≤2 within 2 weeks).
  * grade 4 of any other toxicity (except if return to ≤ G3 within 2 weeks)
  * for all any grade 4 adverse event which lead to treatment discontinuation of more than 7 days
Phase I : to evaluate safety of SBRT | the first 4 weeks (28 days) after the first dose of study treatement for concomitant administration (3X8 Gy of radiotherapy and 3 dosing of immunotherapies)
  Using the following DLTs (DLT are defined by the following events related to study treatments (SBRT and/or tiragolumab, atezolizumab) :
  * grade 3 pneumopathy (except if return to grade ≤2 within 7 days)
  * grade 3 radiation dermatitis (except if return to grade ≤2 within 2 weeks).
  * grade 4 of any other toxicity (except if return to ≤ G3 within 2 weeks)
  * for all any grade 4 adverse event which lead to treatment discontinuation of more than 7 days

SECONDARY OUTCOMES:
Expansion phase : The 6-month progression free survival (PFS) rate after SBRT, atezolizumab and tiragolumab combination. | During 6 months after inclusion
  Evaluation by analysis of PFS. PFS is defined as the time from inclusion to the first occurrence of disease progression, as determined by the investigator according to RECIST v1.1 and iRECIST, or death from any cause, whichever occurs first.It will be evaluated at 6 months.
Expansion cohort : The long term safety of SBRT, atezolizumab and tiragolumab antibodies combination | Throughout the treatment period (24 months)
  Evaluation by analysis of AAE. Will be evaluated with acute and late adverse events (AAEs) according to CTCAE 5.0 Treatment safety evaluation will be based on adverse event (AE) occurrence, the use of concomitant treatments, changes occuring in the course of treatment, observed during physical examination, in the vital signs (arterial pressure, pulse and body temperature), in electrocardiogram (ECG) and biological and clinical examinations (biochemistry, haematology).
Expansion cohort : overall survival (OS) following SBRT, atezolizumab and tiragolumab combination | Until the patient dies
  Evaluation by analysis of Overall survival. Overall survival is defined as the time from inclusion to death to any cause
Expansion cohort : Overall Response rate (ORR) and Non progression rate (NPR) following SBRT, atezolizumab and tiragolumab combination | 18 weeks after inclusion
  Evaluation by analysis of ORR. ORR is evaluated from the first two evaluation scanner images carried out at 8-9 and 16-18 weeks after time from inclusion (CT-scan forecast after the 3rd and the 6th cure) as determined by the investigator according to RECIST v1.1 and iRECIST.
Expansion cohort : The Duration of Response (DOR) and non progression duration (NPD) following SBRT, atezolizumab and tiragolumab combination | Throughout the treatment period (24 months)
  Evaluation by analysis of duration of Response (DOR). DOR is defined as time from documentation of disease complete or partial response to disease progression, defined according to RECISTv1.1 and iRECIST.
  Non Progression duration (NPD) is defined as time from documentation of disease complete response, partial response or stable disease to disease progression, defined according to RECISTv1.1 and iRECIST.
Expansion cohort : To evaluate abscopal effect | Throughout the treatment period (24 months)
  Un-irradiated metastasis volume(s) is evaluated from scanner images

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc (CGFL), Dijon, Bourgogne-Franche-Comté, France

REFERENCES:
- [Derived] Roussot N, Fumet JD, Limagne E, Thibaudin M, Hervieu A, Hennequin A, Zanetta S, Dalens L, Fourrier T, Galland L, Jacob P, Bertaut A, Rederstorff E, Chevalier C, Ghirardi S, Gilbert E, Khoukaz A, Martin E, Nicolet C, Quivrin M, Thibouw D, Vulquin N, Truc G, Rouffiac M, Ghiringhelli F, Mirjolet C. A phase I study of the combination of atezolizumab, tiragolumab, and stereotactic body radiation therapy in patients with metastatic multiorgan cancer. BMC Cancer. 2023 Nov 9;23(1):1080. doi: 10.1186/s12885-023-11534-6. PMID 37946136